CLINICAL TRIAL: NCT05290870
Title: Registry Study on Hydrophilic (HydroSmart) and Hydrophobic (ACUNEX) Intraocular Lenses Manufactured by Teleon Surgical B.V.
Brief Title: Registry Study on Intraocular Lenses Manufactured by Teleon Surgical B.V.
Status: Completed | Type: Observational
Sponsor: Teleon Surgical B.V. (Industry)
Collaborators: MaganaMed GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: PMCF-01-ACX-HS-2022
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Aphakia; Cataract; Clear Lens Exchange; Refractive Lens Exchange
Keywords: Pseudoaphakia
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects implanted with hydrophilic acrylic IOLs: Subjects were implanted with a HydroSmart IOL (FEMTIS, LENTIS or VISIOTIS)
  Interventions: Device: Posterior-chamber intraocular lens
- Subjects implanted with hydrophobic acrylic IOLs: Subjects were implanted with an ACUNEX IOL
  Interventions: Device: Posterior-chamber intraocular lens

INTERVENTIONS:
Device: Posterior-chamber intraocular lens — Implantation of a posterior-chamber intraocular lens to correct aphakia after removal of the crystalline lens

SUMMARY:
This is a retrospective, observational (Registry) study aiming to collect safety and performance data on the use of intraocular lenses (IOLs) manufactured by Teleon Surgical B.V. according to routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Diagnosis of cataract in at least one eye or seeking clear/refractive lens exchange
* Provide consent to retrospective data collection

Exclusion Criteria:

* Patients younger than 18 years
* Patients with congenital primary aphakia or secondary aphakia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone uni- or bilateral extraction of the crystalline lens by means of phacoemulsification or femtosecond laser-assisted cataract surgery with implantation of the subject IOL.
Sampling Method: Non-Probability Sample
Enrollment: 2183 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Visual acuity (uncorrected and/or corrected) | Preoperatively to Month 24
  Monocular visual acuity measured under photopic conditions from preoperative to Month 24 using standard methods (e.g. Snellen Chart 6/6-metre, 1.0 decimal or 0.0 logMAR) at standard distances (4 m for far, 65-80 cm for intermediate and 35-40 cm for near distance), depending on IOL optical design, as follows:
  For monofocal IOLs:
  • Uncorrected and corrected distance visual acuity
  For monofocal toric IOLs:
  * Uncorrected and corrected distance visual acuity
  * Residual astigmatism
  * IOL rotation
  For multifocal IOLs:
  * Uncorrected and corrected distance visual acuity
  * Uncorrected and corrected near visual acuity
  * Uncorrected and corrected intermediate visual acuity, if available
  For multifocal toric IOLs:
  * Uncorrected and corrected distance visual acuity
  * Uncorrected and corrected near visual acuity
  * Uncorrected and corrected intermediate visual acuity, if available
  * Residual astigmatism
  * IOL rotation

SECONDARY OUTCOMES:
Adverse events and adverse device effects | Usual follow-up: 24 Months
Patient and user satisfaction | Month 1
  Satisfaction of the patient with the outcomes of the procedure/medical device Satisfaction of the user with handling of the medical device and patients outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Teleon Surgical B.V., Spankeren, AV, Netherlands

IPD SHARING:
Plan to Share IPD: No